CLINICAL TRIAL: NCT01260103
Title: A Randomized Phase 3 Study of Antineoplastons A10 and AS2-1 vs. Temozolomide in Subjects With Recurrent and / or Progressive Optic Pathway Glioma After Carboplatin or Cisplatin Therapy
Brief Title: Phase 3 Study of ANP Therapy vs. TMZ for Optic Pathway Glioma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawn: study halted prematurely, prior to enrollment of first participant
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRI-BT-54
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Optic Nerve Glioma
Keywords: Optic pathway glioma, recurrent; Optic pathway glioma, progressive; Temozolomide; Temodar; TMZ; Antineoplastons; ANP therapy; Atengenal (A10); Astugenal (AS2-1)
MeSH Terms: conditions — Optic Nerve Glioma; Recurrence | interventions — Temozolomide; antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Temozolomide (TMZ) (Active Comparator): Study subjects receive TMZ for 13 cycles
  Interventions: Drug: Temozolomide
- ANP Therapy (Experimental): Escalating doses of ANP therapy are given daily for 52 weeks.
  Interventions: Drug: ANP Therapy

INTERVENTIONS:
Drug: Temozolomide — Study subjects in a fasting state receive TMZ orally once a day for five consecutive days (days 1 through 5) at a starting dose of 200 mg/m2/day. Treatment cycles are repeated every 28 days following the first daily dose of TMZ from the previous cycle. In the absence of PD or unacceptable toxicity, subjects continue to receive TMZ for a maximum of 13 cycles.
  Other Names: Temodar; TMZ
  Arms: Temozolomide (TMZ)
Drug: ANP Therapy — Escalating doses of ANP therapy are administered for 52 weeks. If the study subject has an OR or maintains SD, ANP therapy is continued.
  Other Names: Antineoplastons; Astengenal (A10); Astugenal (AS2-1)
  Arms: ANP Therapy

SUMMARY:
Primary Objectives

To compare progression free survival (PFS), the time from randomization to progressive disease,in children with optic pathway glioma (OPG) age ≥ 6 months to < 18 years, who receive combination antineoplaston therapy (ANP therapy) vs. temozolomide (TMZ); study subjects will have 1) received prior treatment with carboplatin or cisplatin, which was terminated secondary to toxicity or progression of OPG, or 2) developed recurrence of OPG after completion of carboplatin or cisplatin therapy. PFS data will be censored on the date of the last tumor assessment documenting absence of progression for study subjects:

* Who are alive, on study and are progression-free at the time of the analysis;
* Who discontinue, receive no subsequent therapy and are progression-free at the time of the analysis;
* Who are given/change therapy other than the study treatment prior to observing progression;
* Who discontinued (due to personal preference or toxicity) with a change in therapy, withdrew, or was lost to follow-up;
* For whom documentation of disease progression or death occurs after ≥ 2 consecutive missed tumor assessments.

  * To describe the toxicity profile for ANP therapy vs. TMZ.

Secondary Objectives:

* To compare overall survival (OS) for subjects treated with ANP therapy vs. TMZ;
* To compare disease stabilization rates for subjects treated with ANP therapy vs. TMZ;
* To compare complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD) rates for subjects treated with ANP therapy vs. TMZ.

DETAILED DESCRIPTION:
This is a randomized, phase 3, open-label, multicenter, protocol study in children age ≥ 6 months to < 18 yr., with recurrent and/or progressive OPG who have 1) received prior treatment with carboplatin or cisplatin, which was terminated secondary to toxicity or progression of OPG or 2) developed recurrence of OPG after completion of carboplatin or cisplatin therapy. A total of 158 subjects will be enrolled and randomized equally to one of two therapy groups: ANP therapy (79 subjects) or TMZ (79 subjects). If an average of 4 subjects is enrolled each month, enrollment will be completed in 3 years and 3 months. There will be an additional three years of follow-up.

Children of either gender and from all racial/ethnic groups will be eligible for this protocol study if they meet the criteria outlined in Section 3. Upon determination of eligibility, including the obtaining of an informed consent, study subjects will be randomized to ANP therapy or TMZ. The randomization will be stratified by prior RT (Y/N), hypothalamic involvement (Y/N) and age (< 5 years / ≥ 5 years).

In a group of children treated with TMZ after developing progressive and/or recurrent disease following first-line chemotherapy, a 2-year PFS of 49% and a 4-year PFS of 31% was reported by Gururangan and associates. Based on their results, and assuming an exponential distribution, a least squares estimate of the hazard is 0.333 per year.

For those study subjects, in the BRI Phase 2 study of ANP therapy for OPG, who 1) received prior treatment with carboplatin or cisplatin, which was terminated secondary to toxicity or progression of OPG or 2) developed recurrence of OPG after completion of carboplatin (or cisplatin) therapy, a least squares estimate of the hazard is 0.075 per year. Since the sample size in the Phase 2 study is small and may overstate the effect of ANP therapy in general use, a hazard of 0.167 per year was utilized in determining the sample size for the proposed Phase 3 protocol study, giving a hazard ratio (TMZ:ANP) of 2.0.

The primary efficacy hypothesis of the proposed protocol study is that ANP therapy provides for a significantly better PFS than does TMZ. This protocol study is event-driven (PD or death from any cause), and will be completed after 90 events have occurred. The required sample size in each treatment group is 79.

A log rank test of equality of survival curves, with a 0.05 two-sided significance level, has 90% power to detect the difference in PFS between children treated with ANP therapy vs. children treated with TMZ. Assuming an accrual rate of 4 subjects per month, the accrual period is 3 years and 3 months. There is an additional 3 years of follow-up. A common exponential dropout rate of 0.05 per year is assumed.

This study utilizes an intention-to-treat (ITT) analysis. It is event-driven (PD or death from any cause), and will be completed after 90 events have occurred. All subjects are evaluable for PFS from the time of randomization to the time of PD or death, regardless of therapy group, eligibility, or adequacy of follow-up. All study subjects who receive at least one dose of ANP therapy or TMZ are evaluable for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Children age ≥ 6 months < 18 years are eligible if they have 1) received prior treatment with carboplatin or cisplatin, which was terminated secondary to toxicity or progression of OPG or 2) developed recurrence of OPG after completion of carboplatin or cisplatin therapy.
2. Children with or without prior RT are eligible.
3. Histological confirmation of OPG is required unless the risks of obtaining a diagnostic biopsy are prohibitive.
4. Evidence of OPG (≥ 5 mm), as diagnosed by MRI of the brain, with and without gadolinium contrast, within four weeks of protocol study entry is required. The MRI is interpreted by two independent neuroradiologists. If there is disagreement, a third independent neuroradiologist will adjudicate. Baseline MR spectroscopy (MRS) and positron emission tomography (PET) scan are also performed.
5. Children who are receiving corticosteroids and, for at least one week prior to entry into the protocol study have been on the lowest dose of corticosteroids that preserves optimal neurologic function, are eligible.
6. Children with a life expectancy of > 6 months are eligible.
7. Children ≤ 14 years of age with a Lansky performance status of > 60 are eligible. Children > 14 years of age with a Karnofsky performance status of > 60 are eligible.
8. Children with normal organ and marrow function (as defined below) are eligible.

   * hemoglobin ≥ 10 g/dL
   * leukocytes > 2000/mm3
   * absolute neutrophil count (ANC) >1,500/ mm3
   * serum NA+, K+, BUN within institutional normal limits
   * platelets >75,000/ mm3
   * total bilirubin < 1.5 mg/dL
   * AST(SGOT)/ALT(SGPT) <3 times institutional upper limit of normal (ULN)
   * serum creatinine < 1.5 mg/dL
9. At the recommended therapeutic dose, the effects of ANP therapy on the developing human fetus are unknown. For this reason, women of child-bearing potential who agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to protocol study entry and for the duration of protocol study are eligible. Should a woman become pregnant or suspect she is pregnant while participating in this protocol study, she will inform her treating physician immediately.
10. Children who are able to understand a written informed consent document, and are willing to sign it, are eligible. A subject with a parent or guardian who is able to understand a written informed consent document, and who is willing to sign it on the subject's behalf, is eligible.

Exclusion Criteria:

1. Children receiving prior ANP or TMZ therapy are not eligible.
2. Children with an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled hypertension (> grade 2) or psychiatric illness and/or social situations that would limit compliance with protocol study requirements are not eligible.
3. Children with a history of congestive heart failure, deep venous thrombosis, or other cardiovascular or renal conditions that would contradict administration of high dose intravenous sodium or insertion of a subclavian venous catheter are not eligible.
4. Pregnant women are not eligible because the teratogenic and abortifacient effects of ANP therapy in humans are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to the mother receiving ANP therapy, breastfeeding is discontinued if the mother receives ANP therapy.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 5 years
  PFS will be summarized using tables produced by SAS Proc Lifetest (version 9.2 or later). Standard errors will be computed using the Greenwood formula and 95% confidence intervals produced using the loglog transform. The Log Rank test will be used to compare the two treatment groups with respect to PFS. All tests will be at the two-sided 0.050 significance level.

SECONDARY OUTCOMES:
Safety Analysis | 5 years
  Comparison of the toxicity profile for ANP therapy vs. the toxicity profile for TMZ will be accomplished using the Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R Burzynski, MD, PhD, Study Chair — Burzynski Research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com